CLINICAL TRIAL: NCT06206655
Title: Investigation of Incidence and Proper Diagnostic Method for Adrenal Insufficiency in Liver Cirrhosis Patients
Brief Title: Diagnosis of Adrenal Insufficiency in Liver Cirrhosis Patients
Acronym: DALI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Korea Institute of Science and Technology (Other)
Responsible Party: Principal Investigator, Jung Hee Kim, professor, Seoul National University Hospital
Other Study IDs: 2311-009-1480
Record Dates: First submitted 2024-01-04; First posted 2024-01-16 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Adrenal Insufficiency; Liver Cirrhosis
MeSH Terms: conditions — Adrenal Insufficiency; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum/salivary samples for steroid profiling
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: rapid ACTH stimulation test — Take 2ml blood/saliva sample at baseline. Then, we will inject synacthen 250mcg IV to patients and collect 2ml blood/saliva after 30minutes and 60 minutes.

SUMMARY:
Patients with liver cirrhosis (LC) often exhibit fatigue, poor oral intake, and abdominal discomfort, which are the symptoms that are also shown in subjects with adrenal insufficiency (AI). Controversy exists upon over-diagnosis of adrenal insufficiency in patients with LC, because decreased albumin and/or cortisol binding protein lower total cortisol levels while free cortisol increases/or is preserved. The investigators assumed that measuring salivary cortisol or direct free cortisol using mass-spectrometry would provide a more accurate level of cortisol in LC patients. 50 patients with LC will be recruited and undergo a rapid ACTH stimulation test and their blood/ saliva will be collected and analyzed. The difference between serum free cortisol and total cortisol, as well as between salivary cortisol and total cortisol will be investigated to find the optimal way to diagnose AI in LC patients.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed of liver cirrhosis

Exclusion Criteria:

* pregnant
* history of getting surgery of pituitary resection or adrenalectomy
* patients with diagnosis of pituitary adenoma or adrenal adenoma
* patients take steroid within 3 months
* patients take medication related to synthesis of steroid or cortisol binding protein within 3 months (i.e. ketoconazole, etomidate, sex hormone, oral contraceptive)
* patients take albumin, free frozen plasma, terlipressin, glypressin within 1 month
* patients with acute medical condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients diagnosed of liver cirrhosis without exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Difference between total cortisol, serum free cortisol, and salivary cortisol | baseline, 30 minutes / 60minutes after synacthen injection
  Difference between total cortisol, serum free cortisol, and salivary cortisol

SECONDARY OUTCOMES:
Correlation between serum free cortisol, salivary cortisol and steroid profile | baseline, 30 minutes / 60minutes after synacthen injection
  Correlation between serum free cortisol, salivary cortisol and steroid profile

CONTACTS AND LOCATIONS:
Overall Officials: Junghee Kim, M.D., Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Montagnese S, Middleton B, Mani AR, Skene DJ, Morgan MY. On the origin and the consequences of circadian abnormalities in patients with cirrhosis. Am J Gastroenterol. 2010 Aug;105(8):1773-81. doi: 10.1038/ajg.2010.86. Epub 2010 Mar 23. PMID 20332771
- [Background] Wang S, Cukierman E, Swaim WD, Yamada KM, Baum BJ. Extracellular matrix protein-induced changes in human salivary epithelial cell organization and proliferation on a model biological substratum. Biomaterials. 1999 Jun;20(11):1043-9. doi: 10.1016/s0142-9612(98)00255-5. PMID 10378804
- [Background] Wentworth BJ, Schliep M, Novicoff W, Siragy HM, Geng CX, Henry ZH. Relative adrenal insufficiency in the non-critically ill patient with cirrhosis: A systematic review and meta-analysis. Liver Int. 2023 Mar;43(3):660-672. doi: 10.1111/liv.15473. Epub 2022 Nov 21. PMID 36354293
- [Background] Tripathi PR, Sen Sarma M, Yachha SK, Aggarwal A, Bhatia V, Kumar A, Srivastava A, Poddar U. Relative Adrenal Insufficiency in Decompensated Cirrhotic Children: Does It Affect Outcome? Am J Gastroenterol. 2022 Jan 1;117(1):120-128. doi: 10.14309/ajg.0000000000001486. PMID 34506335
- [Background] Wentworth BJ, Haug RM, Northup PG, Caldwell SH, Henry ZH. Abnormal cholesterol metabolism underlies relative adrenal insufficiency in decompensated cirrhosis. Liver Int. 2021 Aug;41(8):1913-1921. doi: 10.1111/liv.14970. Epub 2021 Jun 8. PMID 34028160